CLINICAL TRIAL: NCT01177748
Title: Stroke Arrhythmia Monitoring Database
Acronym: SAMBA
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Martin Köhrmann, MD, University of Erlangen-Nürnberg Medical School
Other Study IDs: DE-ER-SAMBA
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Acute Stroke
Keywords: Stroke; Cardiac Monitoring
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients on the Stroke Unit

SUMMARY:
Cardiac arrhythmia are frequently observed after stroke. They may on one hand be causative for the stroke mainly in case of atrial fibrillation but on the other hand present severe complications of the stroke. In addition, cardiac comorbidity as well as acute myocardial infarction are frequently found in acute stroke patients. Diagnostics to identify cardiac arrhythmia in the acute phase of stroke care thus have an important role not only for adjusting the correct secondary prevention but also to prevent cardiac complications potentially reducing morbidity and mortality.

The aim of the SAMBA-Study is to systematically assess the prevalence of higher grade arrhythmias after stroke using a standardized reading of 72h telemetric monitoring in the first days after stroke onset. In addition, it evaluates different strategies to identify paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated on the stroke unit
* Patients with telemetric monitoring

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from acute cerebral injury treated on a specialized Stroke Unit
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of high grade cardiac arrhythmia after stroke | 72 hours

SECONDARY OUTCOMES:
Detection of paroxysmal atrial fibrillation by different diagnostic approaches | 72 hours
Cerebral lesion distribution in patients with cardiac arrhythmia | 72 hours
Impact of arrhythmia on clinical outcome and mortality after 90 days | 90 days post stroke

CONTACTS AND LOCATIONS:
Overall Officials: Martin Köhrmann, MD, Principal Investigator — Universityhospital Erlangen; Dept. of Neurology
Locations (1):
- University Hospital Erlangen, Dept. of Neurology, Erlangen, Bavaria, Germany

REFERENCES:
- [Result] Kallmunzer B, Breuer L, Hering C, Raaz-Schrauder D, Kollmar R, Huttner HB, Schwab S, Kohrmann M. A structured reading algorithm improves telemetric detection of atrial fibrillation after acute ischemic stroke. Stroke. 2012 Apr;43(4):994-9. doi: 10.1161/STROKEAHA.111.642199. Epub 2012 Feb 2. PMID 22308240
- [Derived] Kallmunzer B, Breuer L, Kahl N, Bobinger T, Raaz-Schrauder D, Huttner HB, Schwab S, Kohrmann M. Serious cardiac arrhythmias after stroke: incidence, time course, and predictors--a systematic, prospective analysis. Stroke. 2012 Nov;43(11):2892-7. doi: 10.1161/STROKEAHA.112.664318. Epub 2012 Sep 6. PMID 22961962